CLINICAL TRIAL: NCT05248191
Title: Fecal Microbiota Transplant for Postoperative Crohn's Disease
Brief Title: FMT for Postop Crohn's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GI-2022-30546
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; Ileocecal resection; Fecal microbiota transplant; Intestinal microbiota transplant
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial
Who Masked: Participant
Masking Description: Placebo capsules are indistinguishable from study FMT capsules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Capsule fecal microbiota material (cap-FMT) (Experimental): Participants will receive colonoscopy at day 0 and week 8 and receive cap-FMT orally for five days post-colonoscopy. Stool swabs and samples will be collected regularly.
  Interventions: Biological: Capsule fecal microbiota material (cap-FMT)
- Colonoscopic fecal microbiota material (colo-FMT) plus placebo (Active Comparator): Participants will receive colonoscopy at day 0 and week 8 and receive a placebo orally for five days post-colonoscopy. During the first colonoscopy, colo-FMT will be administered. Stool swabs and samples will be collected regularly.
  Interventions: Biological: Colonoscopic fecal microbiota material (colo-FMT)

INTERVENTIONS:
Biological: Capsule fecal microbiota material (cap-FMT) — Cap-FMT consists of Lyophilized FMT administered at 5 x 10^11 bacteria per capsule daily for five days, for a total dose of 2.5 x 10^12 bacteria.
  Arms: Capsule fecal microbiota material (cap-FMT)
Biological: Colonoscopic fecal microbiota material (colo-FMT) — Colo-FMT consists of rehydrated Lyophilized FMT material administered as a single dose of 2.5 x 10^12 bacteria as liquid.
  Arms: Colonoscopic fecal microbiota material (colo-FMT) plus placebo

SUMMARY:
People with Crohn's disease often need surgery. The gut bacteria of people with Crohn's is associated with Crohn's disease coming back after surgery. Fecal microbiota transplant (FMT) after surgery might be a way to prevent Crohn's disease from coming back after surgery.

This study aims to determine if fecal microbiota transplant (FMT) taken by capsules results in the same amount of good bacteria in the guts as FMT by colonoscopy in people with Crohn's disease who have had surgery.

Participants will be randomized to get FMT by capsules or colonoscopy. Colonoscopy with biopsies 8-weeks after the FMT will be used to assess the good bacteria in the gut.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign informed consent form
* Age 18 or older
* English speaking
* Established CD for at least 6-months based on typical clinical, endoscopic, and histopathic evidence.
* Prior ileocecal resection for CD
* Stable medications for 30 days
* Women of reproductive age: Agree to remain abstinent or use effective birth control
* Able and willing to comply with all study procedures

Exclusion Criteria:

* Antibiotic therapy within 15 days
* Probiotic therapy within 15 days
* Adenomatous polyps that have not been removed
* Anticipated antibiotic use over the study period
* Subtotal or total colectomy
* Current ostomy (ileostomy or colonoscopy)
* Anticipated surgical procedure over study period
* Pregnancy
* Severe food allergy
* Diagnosis of end stage liver disease or cirrhosis
* Absolute neutrophil count < 500 cell / uL
* Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-12-25 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Ileal-associated microbiota engraftment | 8 weeks
  Microbiota community of the ileum as sampled by ileal biopsies from colonoscopy. We will use SourceTracker, a Bayesian community-wide software, to assess composition and donor similarity.

CONTACTS AND LOCATIONS:
Overall Officials: Byron Vaughn, MD, MS, Principal Investigator — University of Minnesota Department of Medicine / Gastroenterology, Hepatology, Nutrition
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No